CLINICAL TRIAL: NCT06689020
Title: Effect of Continuous High-frequency Oscillation (CHFO) and Continuous Positive Expiratory Pressure (CPEP) Therapy on Lung RECRUITment Using Electrical Impedance Tomography (EIT) - The PEP-RECRUIT Study
Brief Title: Positive Expiratory Pressure (PEP) and Continuous High-frequency Oscillation (CHFO) on Lung RECRUITment Using Electrical Impedance Tomography (EIT) - The PEP-RECRUIT Study
Acronym: PEP-RECRUIT
Status: Not yet recruiting | Type: Observational
Sponsor: University of Genova (Other)
Collaborators: Denise Battaglini (Unknown)
Responsible Party: Principal Investigator, Lorenzo Ball, Prof., University of Genova
Other Study IDs: PEP-RECRUIT
Record Dates: First submitted 2024-11-11; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Recruitment; Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency | interventions — cholesterylphosphorylethylpyridinium; Therapeutics

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Continuous high-frequency oscillation (CHFO) and continuous positive expiratory pressure (CPEP) therapy — During application of CPEP and CHFO, EIT is monitored.

SUMMARY:
This single-center observational study aims to assess the effects of continuous high-frequency oscillation (CHFO) and continuous positive expiratory pressure (CPEP) therapy on lung recruitment using electrical impedance tomography (EIT) in spontaneously breathing patients admitted to the intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Patients who require pulmonary expansion and airway clearing as per clinical indication
* Patients who provide valid informed consent according to local regulations
* PaO2/FiO2 < 200 mmHg at inclusion
* Patient on the Airway Care Score (ACS) < 7

Exclusion Criteria:

* Refuse to participate
* Age < 18 years
* Hemodynamic instability, defined as systolic arterial pressure < 90 mmHg or mean pressure < 60 mmHg
* Contraindication to using an EIT (i.e., pacemaker or defibrillator)
* Inability to properly position the EIT device for anatomical reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are spontaneously breathing and admitted to the intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 26 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
To assess changes in systemic oxygenation | Immediately before starting treatment (PEP or CHFO), immediately after the end of treatment, at 30 minutes after the end of treatment and at 60 minutes after the end of treatment
  Arterial partial pressure of oxygen (PaO2, mmHg) and PaO2/FiO2 ratio (mmHg)
Changes in lung recruitment using EIT | Immediately before starting treatment (PEP or CHFO), immediately after the end of treatment, at 30 minutes after the end of treatment and at 60 minutes after the end of treatment
  Absolute reduction in the percentage (%) of lung volume collapse assessed with the electrical impedance tomography (EIT)

SECONDARY OUTCOMES:
Mean arterial pressure, mmHg | Immediately before starting treatment (PEP or CHFO), immediately after the end of treatment, at 30 minutes after the end of treatment and at 60 minutes after the end of treatment
  Heart rate as measured by continuous pressure monitoring
Heart rate min-1 | Immediately before starting treatment (PEP or CHFO), immediately after the end of treatment, at 30 minutes after the end of treatment and at 60 minutes after the end of treatment
  Heart rate as measured by continuous electrocardiogram monitoring

CONTACTS AND LOCATIONS:
Locations (1):
- UO Clinica Anestesiologica e Terapia Intensiva, IRCCS Ospedale Policlinico San Martino, Genova, GE, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jonkman AH, Alcala GC, Pavlovsky B, Roca O, Spadaro S, Scaramuzzo G, Chen L, Dianti J, Sousa MLA, Sklar MC, Piraino T, Ge H, Chen GQ, Zhou JX, Li J, Goligher EC, Costa E, Mancebo J, Mauri T, Amato M, Brochard LJ; Pleural Pressure Working Group (PLUG). Lung Recruitment Assessed by Electrical Impedance Tomography (RECRUIT): A Multicenter Study of COVID-19 Acute Respiratory Distress Syndrome. Am J Respir Crit Care Med. 2023 Jul 1;208(1):25-38. doi: 10.1164/rccm.202212-2300OC. PMID 37097986
- [Result] Longhini F, Maugeri J, Andreoni C, Ronco C, Bruni A, Garofalo E, Pelaia C, Cavicchi C, Pintaudi S, Navalesi P. Electrical impedance tomography during spontaneous breathing trials and after extubation in critically ill patients at high risk for extubation failure: a multicenter observational study. Ann Intensive Care. 2019 Aug 13;9(1):88. doi: 10.1186/s13613-019-0565-0. PMID 31410738
- [Result] Battaglini D, Caiffa S, Gasti G, Ciaravolo E, Robba C, Herrmann J, Gerard SE, Bassetti M, Pelosi P, Ball L, On Behalf Of The Gecovid Group. An Experimental Pre-Post Study on the Efficacy of Respiratory Physiotherapy in Severe Critically III COVID-19 Patients. J Clin Med. 2021 May 15;10(10):2139. doi: 10.3390/jcm10102139. PMID 34063429
- [Result] Reychler G, Uribe Rodriguez V, Hickmann CE, Tombal B, Laterre PF, Feyaerts A, Roeseler J. Incentive spirometry and positive expiratory pressure improve ventilation and recruitment in postoperative recovery: A randomized crossover study. Physiother Theory Pract. 2019 Mar;35(3):199-205. doi: 10.1080/09593985.2018.1443185. Epub 2018 Feb 27. PMID 29485340
- [Result] Rowley DD, Malinowski TP, Di Peppe JL, Sharkey RM, Gochenour DU, Enfield KB. A Randomized Controlled Trial Comparing Two Lung Expansion Therapies After Upper Abdominal Surgery. Respir Care. 2019 Oct;64(10):1181-1192. doi: 10.4187/respcare.06812. Epub 2019 May 21. PMID 31113857